CLINICAL TRIAL: NCT05637697
Title: Angelman Syndrome Video Assessment (ASVA) Source Material Study
Acronym: ASVA SMS
Status: Completed | Type: Observational
Sponsor: The Emmes Company, LLC (Industry)
Collaborators: Ionis Pharmaceuticals, Inc. (Industry); Boston Children's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CAS-CAS006
Record Dates: First submitted 2022-08-11; First posted 2022-12-05 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-12

CONDITIONS: Angelman Syndrome
Keywords: Angelman Syndrome
MeSH Terms: conditions — Angelman Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Ambulatory
- Limited Ambulation

SUMMARY:
This is a longitudinal, observational, nonrandomized, fully remote study enrolling approximately 55 participant-caregiver dyads. The study includes no treatments or interventions, and participants will not be asked to change their current treatments. The objective of this study is to gather sufficient source material videos to develop a scoring system for ASVA and to perform preliminary validation of that scoring system.

ELIGIBILITY:
* Caregiver reports that the individual with AS has a laboratory-confirmed diagnosis of Angelman syndrome
* Individual with AS is at least 1 year old
* Caregiver is willing and able to provide informed consent for themselves and oversee study participation
* Caregiver or legal guardian is willing to provide informed consent on behalf of the individual with AS
* Caregiver is comfortable reading and speaking in English
* Caregiver has access to a smartphone or tablet that is compatible with the study app OR caregiver has internet access and is willing to use a wi-fi only device to record and upload videos

NT-Caregiver dyads will be eligible for inclusion if the:

* Neurotypical individual is between 1 and 8 years of age
* Caregiver is willing and able to provide informed consent and oversee study participation and NT individual is willing and able to provide assent, as applicable
* Caregiver is comfortable reading and speaking in English
* Caregiver has access to a smartphone or tablet that is compatible with the study app OR caregiver has internet access and is willing to use a wi-fi only device to record and upload videos Participant-Caregiver dyads will be excluded from the study only if they do not meet the inclusion criteria above.

Min Age: 1 Year | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: 40 participants with Angelman Syndrome (AS) and their caregivers (AS-caregiver dyads) and up to 15 neurotypically (NT) developing children and their caregivers (NT-caregiver dyads) for a total of up to 55 participant-caregiver dyads. AS-caregiver dyads will be recruited for this study through referrals from collaborators and advocacy groups as well as through direct marketing via social media.
Sampling Method: Non-Probability Sample
Enrollment: 73 (Actual)
Dates: Start 2021-08-31 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
Source material collection, Baseline | Baseline
  The objective of this study is to gather sufficient source material videos to develop a scoring system for ASVA and to perform preliminary validation of that scoring system.
Source material collection, Week 12 | Week 12
  The objective of this study is to gather sufficient source material videos to develop a scoring system for ASVA and to perform preliminary validation of that scoring system.

CONTACTS AND LOCATIONS:
Overall Officials: Mindy Leffler, Principal Investigator — Casimir
Locations (1):
- Casimir, Kingston, Massachusetts, United States

DOCUMENTS (1):
  • Study Protocol (2022-05-02): https://cdn.clinicaltrials.gov/large-docs/97/NCT05637697/Prot_000.pdf